CLINICAL TRIAL: NCT05955456
Title: Detecting EARLY Heart Failure in Greater Manchester (EARLY-HF)
Brief Title: Detecting EARLY Heart Failure in Greater Manchester
Acronym: EARLY-HF
Status: Recruiting | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: B01899
Record Dates: First submitted 2023-07-13; First posted 2023-07-21 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants in primary care with risk factors for heart failure
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention is applied to participants. The risk calculator score is not released to the participants or care providers. Participants are followed up for risk calculator accuracy and recalibration.

SUMMARY:
Heart failure represents a growing public health problem within the UK and particularly within the North West of England. A major challenge is that heart failure is currently diagnosed too late.

The researchers have previously developed a risk calculator that accurately identifies individuals at risk of heart failure admission or death before they have developed heart failure.

Most risk calculators are never implemented into clinical practice. The researchers will l perform a pilot study to evaluate the risk calculator within primary care in Greater Manchester.

DETAILED DESCRIPTION:
The researchers have previously developed and externally validated a novel multimodal risk calculator that accurately identifies individuals at-risk of heart failure admission or death before they have developed heart failure. This risk calculator includes key co-morbidities, circulating biomarkers and cardiac magnetic resonance imaging (CMR) measurements of cardiac structure and function. It identifies those individuals at highest risk of developing heart failure and therefore those who may most benefit from targeted cardiometabolic therapeutics in the future.

The researchers will l perform a pilot study to evaluate the risk calculator within primary care in Greater Manchester. A qualitative and quantitative assessment of risk calculator uptake will be performed within local GP practices and primary care populations. The research team will determine how effectively they can recruit participants from socioeconomically deprived and ethnically diverse backgrounds. A preliminary analysis will be performed to determine risk calculator accuracy within a prospective primary care cohort, and dynamically refine the model aiming to improve performance. The study will also involve conducting an initial cost effectiveness analysis to determine the real-world economic impact of model implementation.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Aged 50 and over
* Two or more of the following conditions: type 2 diabetes, chronic obstructive pulmonary disease, ischaemic heart disease, atrial fibrillation, hypertension, chronic kidney disease stage 3, body mass index ≥ 30 kg/m2

Exclusion Criteria:

* Established diagnosis of one or more of the following: heart failure, cardiomyopathy, moderate or severe valvular heart disease, congenital heart disease, heart transplant, idiopathic, heritable or drug-induced pulmonary arterial hypertension, any medical condition, which in the opinion of the Investigator, may place the patient at higher risk from his/her participation in the study, or is likely to prevent the patient from complying with the requirements of the study or completing the study.
* Contraindication to cardiovascular magnetic resonance (CMR) scanning, including pacemaker, defibrillator, intraocular metal, intracranial aneurysm clips, severe claustrophobia, estimated glomerular filtration rate < 30 ml/min/1.73m2, previous severe allergic reaction or anaphylaxis to gadolinium-based contrast agent, pregnancy or breastfeeding.

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Primary care population with risk factors for heart failure
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2030-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Preliminary measures of risk calculator validation and accuracy in Greater Manchester | 5 years
  Risk calculator will predict incident heart failure, first heart failure hospitalisation, cardiovascular death and all cause death

SECONDARY OUTCOMES:
Qualitative measures of primary care uptake and engagement | 5 years
  Number of participant identification sites, methods of participant identification, proportion of eligible participants contacted and recruited
Proportion of participants recruited from socioeconomically deprived and ethnically diverse backgrounds | 5 years
  Ability to recruit participants from socioeconomically deprived and ethnically diverse backgrounds within Greater Manchester
Measures of prognostic model calibration and discrimination in a primary care population | 5 years
  Examples include calibration slope, intercept and Harrell's C statistic
Measures of prognostic model optimisation and accuracy with iterative variable inclusion or exclusion | 5 years
  Assess variable inclusion and exclusion using stepwise model selection and Wald statistic
Causal statistical analysis to determine effect of hypothetical interventions | 5 years
  Mediation analysis to determine causative effects of hypothetical interventions
Measures of cost effectiveness of the model in Greater Manchester | 5 years
  Examples include decision curve analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided